CLINICAL TRIAL: NCT00751751
Title: Comparison of the Efficacy of Olmesartan Medoxomil Versus Losartan on Diastolic Blood Pressure in Elderly and Very Elderly Patients With Essential Hypertension.
Brief Title: Olmesartan Medoxomil Versus Losartan in Elderly and Very Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Petra Laeis, Ph.D., Daiichi Sankyo Europe, GmbH
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SE-866/36
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Olmesartan Medoxomil; Hydrochlorothiazide; Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): oral olmesartan medoxomil tablets 20 or 40 mg taken once daily for 52 weeks + hydrochlorothiazide tablets 12.5 or 25 mg , if needed to control BP after 12 weeks
  Interventions: Drug: olmesartan medoxomil + hydrochlorothiazide, if necessary
- 2 (Active Comparator): oral losartan capsules, 50 or 100 mg taken once daily for 52 weeks + 12.5 or 25 mg oral hydrochlorothiazide tables, after 12 weeks, if needed to control BP.
  Interventions: Drug: losartan + hydrochlorothiazide, if necessary

INTERVENTIONS:
Drug: olmesartan medoxomil + hydrochlorothiazide, if necessary — oral olmesartan medoxomil tablets taken once daily for 52 weeks + oral hydrochlorothiazide tablets, once daily, after 12 weeks if needed to control BP
  Arms: 1
Drug: losartan + hydrochlorothiazide, if necessary — oral losartan capsules, 50 or 100 mg taken once daily for 52 weeks + 12.5 or 25 mg oral hydrochlorothiazide tablets, after 12 weeks, if needed to control BP.
  Arms: 2

SUMMARY:
To assess the efficacy of individually optimized doses of olmesartan medoxomil compared to losartan in elderly and very elderly patients with essential hypertension. The study hypothesis is non-inferiority of olmesartan medoxomil compared to losartan in lowering mean sitting diastolic blood pressure after 12 weeks of treatment compared to baseline. The study duration is up to 60 weeks, including a 52-week treatment period. After 12 weeks of treatment hydrochlorothiazide may be added to control blood pressure. Efficacy and safety measurements are carried out at up to 18 visits during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Mean sitting diastolic BP = 100-114 mmHg and mean sitting systolic BP >=150 mm HG

Exclusion Criteria:

* Secondary hypertension
* Malignant hypertension
* Severe heart failure (NYHA III-IV)
* History or evidence of renal disease
* Recent history of myocardial infarction
* Hypersensitivity to study drugs
* History of drug or alcohol abuse

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 441 (Actual)
Dates: Start 2003-06; Primary Completion 2005-04 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change in mean sitting diastolic blood pressure assessed by conventional BP measurements | 12 weeks

SECONDARY OUTCOMES:
Change in mean sitting diastolic BP assessed by conventional BP measurements | after 1, 2, 4, 8, 16, 20, 28, 36, 44, and 52 weeks
Change in mean standing diastolic BP, mean sitting systolic BP and mean standing systolic BP | after 1, 2, 4, 8, 12, 16, 20, 28, 36, 44, and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter U Witte, MD, Ph.D., Principal Investigator — IMFORM GmbH
Locations (1):
- Darmstadt, Germany